CLINICAL TRIAL: NCT06508710
Title: Early Efficacy of Ketamine Compared With Placebo as Adjunctive Therapy With Venlafaxine in Severely Unipolar Depressed Inpatients
Brief Title: Early Effects of Ketamine vs Placebo With Venlafaxine in Severe Depression Patients
Acronym: MOODBOOSTER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP220668; 2023-506597-12-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-15; First posted 2024-07-18 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2024-12

CONDITIONS: Major Depressive Episode
Keywords: depression; ketamine; synaptogenesis
MeSH Terms: conditions — Depression | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine Group (Experimental): The patient will receive 3 doses of intravenous ketamine (0,50mg/kg) in addition to the usual venlafaxine treatment
  Interventions: Drug: Ketamine
- Placebo group (Placebo Comparator): The patient will receive 3 doses of intravenous placebo (50mL of NaCl 9‰) in addition to the usual venlafaxine treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — Patients randomized in this group will receive an intravenous ketamine in addition to venlafaxine for one week (on Days 1, 4 and 7)
  Other Names: Ketamine+Venlafaxine
  Arms: Ketamine Group
Drug: Placebo — Patients randomized in this group will receive an intravenous placebo in addition to venlafaxine for one week (on Days 1, 4 and 7)
  Other Names: Placebo+Venlafaxine
  Arms: Placebo group

SUMMARY:
Unipolar major depressive disorder is the leading cause of disability worldwide. The most commonly used treatments for major depressive episodes (MDE) are antidepressant medications. However, they have limited efficacy and their onset of action is long, ranging between 2 to 6 weeks. During this period, hospitalization can become necessary, especially for severe MDE. It is crucial to improve the early effectiveness of treatments for these patients in order to alleviate their suffering, limit complications (suicidal risk), and reduce hospitalization durations (approximately 1000 euros per day). The efficacy of intravenous ketamine has been demonstrated in pharmaco-resistant depression but remains to be proven in non-pharmaco-resistant severe MDE. Additionally, PET imaging using [11C]UCB-J, which allows the in vivo study of synaptic density in the human brain, has shown significant decreases in synaptic density in unipolar patients with severe MDE. Furthermore, a single ketamine infusion was found to enhance synaptogenesis

ELIGIBILITY:
Inclusion Criteria:

* Current MDE in the context of unipolar major depressive disorder (DSM-5 criteria), hospitalized (open care) for this episode, with a minimum HDRS score of 24 and in the context of an indication for the introduction of venlafaxine treatment.
* Patient aged between 18 and 65.
* Signed free and informed consent
* Membership of a social security scheme
* For women of childbearing age, effective contraception throughout study participation.* (*Combined hormonal contraception (containing estrogen and progestin) associated with ovulation inhibition: (oral, intravaginal, transdermal), Progestin-only hormonal contraception associated with ovulation inhibition: (oral, injectable, implantable), Intrauterine device (IUD), Hormonal intrauterine system (IUS), Bilateral tubal occlusion, Vasectomized partner, Sexual abstinence.)

Exclusion Criteria:

* Criteria relating to associated pathologies entailing particular risks: pharmaco-resistant CDE (failure of at least two properly conducted treatments with two different antidepressant treatment classes), CDE with psychotic features, psychotic disorder, bipolar disorder, current (<1 month) substance use disorder (excluding tobacco).
* Liver impairment (AST and/or ALT > 3 ULN, PAL and/or GGT and/or bilirubin > 2 ULN).
* Severe renal insufficiency (GFR <30ml/min with Cockcroft's formula).
* Bradycardia less than 55 beats per minute.
* Contraindication to ketamine : Hypersensitivity to active substance or excipients, comatose state, central nervous system (CNS) depression, Parkinson's disease, Lewy body dementia, progressive supranuclear palsy, known prolongation of the QTc interval (>450ms for men and >470ms for women) or congenital long QT syndrome, recent acute myocardial infarction, uncompensated heart failure, history of ventricular arrhythmias or torsades de pointes, uncorrected hypokalemia (K+ < 3. 5 mmol/l), epilepsy, uncontrolled hypertension, porphyria, history of stroke (CVA), intracranial hypertension.
* Contraindication to venlafaxine (hypersensitivity to venlafaxine or excipients, are hereditary conditions of fructose intolerance, glucose-galactose malabsorption syndrome, or sucrase-isomaltase deficiency, unstable hypertension, no indication for venlafaxine treatment in clinician's opinion due to ineffectiveness or tolerability of previous venlafaxine treatment).
* Current or previous treatment with venlafaxine or ketamine in the month prior to study inclusion.
* Need to maintain another antidepressant, MAOI, Millepertuis or benzodiazepines (cyamemazine is permitted). Or potential drug interactions in case of recent cessation of these treatments (based on the Summary of Product Characteristics (SmPC) of the respective medication(s) and their half-life).
* Any other unspecified reason (clinically significant illness or anomaly) which, in the opinion of the investigator or the sponsor, could compromise the safety of the participant.
* Pregnant or breast-feeding patients (women of childbearing potential must have a negative urine or blood test for human chorionic gonadotropin prior to trial entry). Planned pregnancy within three months of enrolment
* Adult under guardianship, curatorship or safeguard of justice
* Participating in other interventional research involving the human body or within the exclusion period following previous research involving the human body, if applicable.
* Social insurance

Additional criteria for inclusion in the ancillary study :

- Contraindications to [11C]UCB-J PET-MRI

1. Absolute contraindications: Pacemaker or neurosensorial stimulator or implantable defibrillator; clip on a brain aneurysm or vascular malformation; intraocular or intracerebral ferromagnetic foreign body; prostheses or objects or mobile ferromagnetic metal fragments; cochlear implants; peripheral stimulator; neurosurgical ventriculoperitoneal shunt valves; automated injection device such as insulin pump, glucose sensor; permanent eyelid or lip makeup; non-removable piercing; claustrophobia.
2. Relative contraindications: Dental prostheses and orthodontic material; certain intrauterine devices; certain tattoos; certain transdermal patch implants; certain metal implants far from the examined area. (The investigator physician and/or radiology operator will always conduct a precise questionnaire before the examination to ensure perfect safety and absence of MRI danger)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
the early efficacy on depressive symptomatology | at day 0 and day 7
  Evolution of the total score of the Hamilton Depression Rating Scale (HDRS 17 items: scale items are rated from 0 to 2 or from 0 to 4 and the score ranges from 0 to 52) after 7 days of treatment by venlafaxine The HDRS scale will be assessed by a senior psychiatrist or psychologist trained in administering the scales, following a psychiatric interview

SECONDARY OUTCOMES:
The efficacy of ketamine on HDRS overall score | at day 1,4,7,14, 28 and 42 following the initiation of treatment by venlafaxine
  To compare the efficacy of ketamine as adjunctive therapy, after the early adjunctive treatment phase, and placebo, by assessing changes in overall score obtained on the HDRS 17-items.
The efficacy of Ketamine on HDRS response rate | at day 1,4,7,14, 28 and 42 following the initiation of treatment by venlafaxine
  To compare the efficacy of ketamine as adjunctive therapy, after the early adjunctive treatment phase, and placebo, by assessing HDRS response rate (improvement of 50% or more in the overall HDRS score) between groups
The efficacy of Ketamine on HDRS remission rate | To compare the efficacy of ketamine as adjunctive therapy, after the early adjunctive treatment phase, and placebo, by assessing remission rate (HDRS 17 items ≤ 7) between groups
  at day 1,4,7,14, 28 and 42 following the initiation of treatment by venlafaxine
The efficacy of ketamine on BDI overall score | at day 1,4,7,14, 28 and 42 following the initiation of treatment by venlafaxine
  To compare the efficacy of ketamine as adjunctive therapy, after the early adjunctive treatment phase, and placebo, by assessing changes in overall score obtained on the short form of the Beck Depression Inventory (BDI)
The efficacy of ketamine on CGI scale | at day 1,4,7,14, 28 and 42 following the initiation of treatment by venlafaxine
  To compare the efficacy of ketamine as adjunctive therapy, after the early adjunctive treatment phase, and placebo, by assessing changes in Clinical Global Impression (CGI) scale
Duration of hospitalization | 42 days
  Evaluate whether ketamine as adjunctive therapy reduces the length of hospital stay, noting the number of days spent in hospital (including re-hospitalization) The discharge from hospitalization will be decided by the treatment-blinded clinician responsible for the patient
Reduction of suicidal ideation | at day 0 and day 7
  Evaluate whether adjunctive ketamine reduces early suicidal ideation, by assessement of overall Columbia-Suicide Severity Rating Scale (C-SSRS) score, after 7 days of treatment by venlafaxine
Clinical improvement on HDRS overall score | at day 7, 14, 28 and 42
  Evaluate whether ultra-early improvement (at D1 or D4 of treatment by venlafaxine) predicts clinical improvement at D7, D14, D28 and D42 by tracking changes in overall score obtained on the 17-item Hamilton Depression Rating Scale (HDRS)
Clinical improvement on HDRS response rate | at day 7, 14, 28 and 42
  Evaluate whether ultra-early improvement (at D1 or D4 of treatment by venlafaxine) predicts clinical improvement at D7, D14, D28 and D42 by tracking HDRS response rate (improvement of 50% or more in the overall HDRS score)
Clinical improvement on HDRS remission rate | at day 7, 14, 28 and 42
  Evaluate whether ultra-early improvement (at D1 or D4 of treatment by venlafaxine) predicts clinical improvement at D7, D14, D28 and D42 by tracking remission rate (HDRS 17 items ≤ 7)
Clinical improvement on BDI overall score | at day 7, 14, 28 and 42
  Evaluate whether ultra-early improvement (at D1 or D4 of treatment by venlafaxine) predicts clinical improvement at D7, D14, D28 and D42 by tracking changes in overall score obtained on the short form of the Beck Depression Inventory (BDI)
Clinical improvement on CGI scale | at day 7, 14, 28 and 42
  Evaluate whether ultra-early improvement (at D1 or D4 of treatment by venlafaxine) predicts clinical improvement at D7, D14, D28 and D42 by tracking changes in Clinical Global Impression (CGI) scale
Tolerance on blood pressure | Day 1, 4, 7
  Tolerance will be assessed according to CTCAE grade (version 5.0), with special monitoring of the effects of ketamine during and up to 40 minutes post-infusion of treatment or placebo on blood pressure
Tolerance on heart rate | Day 1, 4, 7
  Tolerance will be assessed according to CTCAE grade (version 5.0), with special monitoring of the effects of ketamine during and up to 40 minutes after infusion of treatment or placebo on heart rate.
Tolerance on respiratory rate | Day 1, 4, 7
  Tolerance will be assessed according to CTCAE grade (version 5.0), with special monitoring of the effects of ketamine during and up to 40 minutes after infusion of treatment or placebo on respiratory rate
Tolerance on nausea and vomiting | Day 1, 4, 7
  Tolerance will be assessed according to CTCAE grade (version 5.0), with special monitoring of the effects of ketamine during and up to 40 minutes after infusion of treatment or placebo on nausea/vomiting
Tolerance on dissociation | Day 1, 4, 7
  Tolerance will be assessed according to CTCAE grade (version 5.0), with special monitoring of the effects of ketamine during and up to 40 minutes after infusion of treatment or placebo on dissociation
Tolerance on headaches | Day 1, 4, 7
  Tolerance will be assessed according to CTCAE grade (version 5.0), with special monitoring of the effects of ketamine during and up to 40 minutes after infusion of treatment or placebo on headaches
The consumption of anxiolytic treatments | During all the study
  cumulative consumption in mg of cyamemazine will be recorded over the entire study period
Biomarkers | Day 1 and 14
  Identify biomarkers predictive or associated with the efficacy of venlafaxine associated with ketamine

OTHER OUTCOMES:
Synaptic density variation in the whole brain | Day 0 and 14
  Within-subject variation in synaptic density between day 0 and day 14 following treatment initiation of venlafaxine, estimated by measuring the rate of [11C]UCB-J binding to SV2A proteins by PET-MRI in the whole brain
synaptic density variation in the cingulate cortex | Day 0 and 14
  Within-subject variation in synaptic density between day 0 and day 14 following treatment initiation of venlafaxine, estimated by measuring the rate of [11C]UCB-J binding to SV2A proteins by PET-MRI in the cingulate cortex
synaptic density variation in the prefrontal cortex | Day 0 and 14
  Within-subject variation in synaptic density between day 0 and day 14 following treatment initiation of venlafaxine, estimated by measuring the rate of [11C]UCB-J binding to SV2A proteins by PET-MRI in the prefrontal cortex
synaptic density variation in the hippocampus | Day 0 and 14
  Within-subject variation in synaptic density between day 0 and day 14 following treatment initiation of venlafaxine, estimated by measuring the rate of [11C]UCB-J binding to SV2A proteins by PET-MRI in the hippocampus
Relationship between ketamine efficacy and synaptogenesis | Day 0 and 14
  Correlation between changes in the HDRS scale and within-subject variation in synaptic density between day 0 and day 14 following treatment initiation of venlafaxine.

CONTACTS AND LOCATIONS:
Overall Officials: Romain COLLE, Principal Investigator — Service Hospitalo-Universitaire de Psychiatrie - Hôpital Bicêtre
Locations (4):
- France (4):
  - Psychiatry unit, Le Kremlin-Bicêtre, France
  - EPS Barthélémy Durand, Étampes
  - Bicetre Hospital - CRC, Le Kremlin-Bicêtre
  - CEA/SHFJ, Orsay